CLINICAL TRIAL: NCT05590884
Title: Gadopiclenol Pharmacokinetics, Safety and Efficacy in Pediatric Patients < 2 Years of Age
Brief Title: Gadopiclenol Pharmacokinetics, Safety and Efficacy in Children < 2 Years of Age
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Guerbet (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: GDX-44-015
Record Dates: First submitted 2022-10-18; First posted 2022-10-21 (Actual); Results first posted 2025-10-28 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Central Nervous System Diseases; Pediatric Disorder; Body Indication
MeSH Terms: conditions — Central Nervous System Diseases | interventions — gadopiclenol

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Age Group 1: patients aged 3 to 23 months (Experimental): One Investigational Medicinal Product (IMP) dose of 0.05 mmol/kg will be injected in all patients.
  Interventions: Drug: Gadopiclenol
- Age Group 2: patients aged 28 days to less than 3 months (Experimental): One Investigational Medicinal Product (IMP) dose of 0.05 mmol/kg will be injected in all patients.
  Interventions: Drug: Gadopiclenol
- Age Group 3: patients aged from birth to 27 days (term newborns) (Experimental): One Investigational Medicinal Product (IMP) dose of 0.05 mmol/kg will be injected in all patients.
  Interventions: Drug: Gadopiclenol

INTERVENTIONS:
Drug: Gadopiclenol — Patients will receive a single dose of gadopiclenol calculated according to their BW on the day of MRI examination. Gadopiclenol will be administered at a dose of 0.05 mmol/kg BW (0.1 mL/kg BW).
  Other Names: Elucirem

SUMMARY:
This Phase II open-label, uncontrolled, multicenter trial is designed to investigate the pharmacokinetic (PK) profile of gadopiclenol in plasma, in pediatric patients aged up to 23 months inclusive (term neonates or preterm infants after the neonatal period), using a population PK approach.

Primary objective is to evaluate the PK profile of gadopiclenol in plasma following single intravenous injection of 0.05 mmol/kg body weight (BW) in pediatric population aged up to 23 months (inclusive) scheduled for a contrast-enhanced MRI examination of any body region including central nervous system (CNS).

DETAILED DESCRIPTION:
Three age groups are defined:

* Group 1: patients aged 3 to 23 months (inclusive)
* Group 2: patients aged 28 days to less than 3 months;
* Group 3: patients aged from birth to 27 days (term newborns).

At study set-up, the inclusions started with the oldest patients in group 1 and using an age-down staggered approach.

The decision to start the inclusions in group 2 was taken by the Trial Safety Review Board based on safety assessment over one-day period after injection of the first 13 patients in group 1.

According to the protocol version 4 (amendments 2 & 3), the age-down staggered approach was discontinued to allow the inclusions in Group 3 (patients aged from birth to 27 days), simultaneously to inclusions in group 1 and group 2.

A total of 3 blood samples per patient were taken post-injection for PK analysis.

ELIGIBILITY:
Main Inclusion Criteria:

1. Female or male pediatric patient aged from birth to 23 months of age inclusive (term neonates for all age groups or preterm infants after the neonatal period for groups 1 or 2). The neonatal period for preterm newborns is defined as the day of birth through the expected date of delivery plus 27 days. Term is defined as ≥37 completed weeks of amenorrhea,
2. Patient with known or highly suspected abnormalities/ lesion(s), scheduled to undergo contrast-enhanced MRI of any body region including CNS [...]

Main Exclusion Criteria:

1. Patient planned for treatment or procedure (e.g. surgery) that would prevent from obtaining the required blood samples or performing other trial procedures between the screening visit and up to one day after gadopiclenol administration,
2. Patient undergoing treatment or procedure (e.g., diuretics, clinically significant blood loss or blood transfusion) preceding or subsequent to gadopiclenol administration that would alter gadopiclenol pharmacokinetic parameters,
3. Patient with acute or chronic renal insufficiency defined as estimated Glomerular Filtration Rate (eGFR) out of age-adjusted normal value calculated based on bedside Schwartz equation, [...]

9. Patient undergoing a change in chemotherapy (product or dosage) within one day prior to or one day after gadopiclenol administration, 10. Patient who received or will receive any other contrast agent for CT and/or MRI within one week prior to or one week after gadopiclenol administration, 11. Patient with contraindication for MRI such as iron metal implants (e.g., aneurysm clips, pacemaker), 12. Patient with history of anaphylactoid or anaphylactic reaction to any allergen including drugs and contrast agents [...]

Max Age: 23 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2022-09-21 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donna R Roberts, MD, Principal Investigator — Medical University of South Carolina, Division of Neuroradiology
Locations (11):
- United States (2):
  - Cincinnatti Childrens Hospital, Cincinnati, Ohio
  - Medical University of South Carolina, Charleston, South Carolina
- Hungary (3):
  - Semmelweis Egyetem, Budapest
  - Országos Idegtudományi Intézet, Budapest
  - University of Debrecen Clinical Center Pediatric Department, Debrecen
- Poland (6):
  - Szpital Uniwersytecki nr 1 im. dr Antoniego Jurasza, Bydgoszcz
  - Instytut Centrum Zdrowia Matki Polki, Lodz
  - Uniwersytecki Szpital Dzieciecy, Lublin
  - Kliniczny Szpital Wojewodzki Nr 2 im. Sw. Jadwigi Krolowej, Rzeszów
  - Uniwersyteckie Centrum Kliniczne Warszawskiego, Warsaw
  - Instytut "Pomnik - Centrum Zdrowia Dziecka", Warsaw

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Age Group 1: Patients Aged 3 to 23 Months; Age Group 2: Patients Aged 28 Days to Less Than 3 Months; Age Group 3: Patients Aged From Birth to 27 Days (Term Newborns): One Investigational Medicinal Product (IMP) dose of 0.05 mmol/kg was injected in all patients.
  Gadopiclenol: Patients received a single dose of gadopiclenol calculated according to their BW on the day of MRI examination. Gadopiclenol was administered at a dose of 0.05 mmol/kg BW (0.1 mL/kg BW).
Period: Overall Study
Arm/Group | Age Group 1: Patients Aged 3 to 23 Months | Age Group 2: Patients Aged 28 Days to Less Than 3 Months | Age Group 3: Patients Aged From Birth to 27 Days (Term Newborns)
Started | 33 | 2 | 1
Completed | 32 | 2 | 1
Not Completed | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline analysis population included 36 patients who received one injection of gadopiclenol (safety set): 33 patients aged 3 to 23 months, 2 aged 28 days to less than 3 months and 1 patient aged 0-27 days.
Groups:
- Total: Total of all reporting groups
Arm/Group | Age Group 1: Patients Aged 3 to 23 Months | Age Group 2: Patients Aged 28 Days to Less Than 3 Months | Age Group 3: Patients Aged From Birth to 27 Days (Term Newborns) | Total
Number analyzed (Participants) | 33 | 2 | 1 | 36
Age, Continuous [Mean (Standard Deviation); unit: months] | 13.11 (6.22) | 1.94 (0.14) | 0.8 (NA) — only one participant | 12.15 (6.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 1 | 0 | 18
  Male | 16 | 1 | 1 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 32 | 2 | 1 | 35
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 33 | 2 | 1 | 36
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Hungary | 10 | 1 | 1 | 12
  United States | 4 | 1 | 0 | 5
  Poland | 19 | 0 | 0 | 19
Weight [Mean (Standard Deviation); unit: kilogram] | 9.40 (2.18) | 5.10 (0.28) | 4.50 (NA) — only one patient | 9.03 (2.44)

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve (AUCinf)
Description: Exposure parameter by age group predicted from the final model in participants with normal renal function receiving gadopiclenol at a dose of 0.05 mmol/kg
Time Frame: A total of 3 blood samples per patient were collected post-injection of gadopiclenol for PK analysis, one within each window (10-60 minutes, 2-4 hours and 6-8 hours)
Population: Among the 36 patients who received an injection of gadopiclenol for MRI (Safety Set), the patient aged 0-27 days was excluded from the Per Protocol Set, due to a major deviation impacting the popPK model, therefore 35 patients were included in the population PK analysis including 33 patients aged 3-23 months and 2 patients aged 28-89 days.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h.mg/L
Groups:
- Age Group 1: Patients Aged 3 to 23 Months: Patients aged 3-23 months who underwent a contrast-enhanced MRI examination of any body region including central nervous system (CNS cohort) or vessels (Blood vessel cohort) or others region (Body cohort) with a single injection of gadopiclenol at a dose of 0.05 mmol/kg body weight (0.1 mL/kg body weight).
- Age Group 2: Patients Aged 28 Days to Less Than 3 Months: Patients aged 28-89 days who underwent a contrast-enhanced MRI examination of any body region including central nervous system (CNS cohort) or vessels (Blood vessel cohort) or others region (Body cohort) with a single injection of gadopiclenol at a dose of 0.05 mmol/kg body weight (0.1 mL/kg body weight).
- Age Group 3: Patients Aged From Birth to 27 Days (Term Newborns): Patients aged from birth to 27 days who underwent a contrast-enhanced MRI examination of any body region including central nervous system (CNS cohort) or vessels (Blood vessel cohort) or others region (Body cohort) with a single injection of gadopiclenol at a dose of 0.05 mmol/kg body weight (0.1 mL/kg body weight).
Arm/Group | Age Group 1: Patients Aged 3 to 23 Months | Age Group 2: Patients Aged 28 Days to Less Than 3 Months | Age Group 3: Patients Aged From Birth to 27 Days (Term Newborns)
Number analyzed (Participants) | 33 | 2 | 0
h.mg/L | 392.3 (27.6) | 493.3 (9.9) |

2. Primary Outcome: Elimination Half-life (t1/2α)
Description: as for outcome 1
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h
Arm/Group | Age Group 1: Patients Aged 3 to 23 Months | Age Group 2: Patients Aged 28 Days to Less Than 3 Months | Age Group 3: Patients Aged From Birth to 27 Days (Term Newborns)
Number analyzed (Participants) | 33 | 2 | 0
h | 0.3 (30.3) | 0.3 (30.3) |

3. Primary Outcome: Terminal Half-life (t1/2β)
Description: as for outcome 1
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h
Arm/Group | Age Group 1: Patients Aged 3 to 23 Months | Age Group 2: Patients Aged 28 Days to Less Than 3 Months | Age Group 3: Patients Aged From Birth to 27 Days (Term Newborns)
Number analyzed (Participants) | 33 | 2 | 0
h | 1.5 (21.4) | 2.1 (8.4) |

4. Primary Outcome: Gadopiclenol Concentrations 10 Min Post-injection (C10 Min)
Description: as for outcome 1
Time Frame: blood sample collection 10 minutes post-injection of gadopiclenol for analysis
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg/L
Arm/Group | Age Group 1: Patients Aged 3 to 23 Months | Age Group 2: Patients Aged 28 Days to Less Than 3 Months | Age Group 3: Patients Aged From Birth to 27 Days (Term Newborns)
Number analyzed (Participants) | 33 | 2 | 0
mg/L | 226.8 (15.8) | 190.4 (16.2) |

5. Primary Outcome: Gadopiclenol Concentration 20 Min Post-injection (C20 Min)
Description: as for outcome 1
Time Frame: blood sample collection 20 minutes post-injection of gadopiclenol
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg/L
Arm/Group | Age Group 1: Patients Aged 3 to 23 Months | Age Group 2: Patients Aged 28 Days to Less Than 3 Months | Age Group 3: Patients Aged From Birth to 27 Days (Term Newborns)
Number analyzed (Participants) | 33 | 2 | 0
mg/L | 161.5 (17.2) | 149.8 (13.4) |

6. Primary Outcome: Gadopiclenol Concentrations 30 Min Post-injection (C30 Min)
Description: as for outcome 1
Time Frame: blood sample collection 30 minutes post-injection of gadopiclenol
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg/L
Arm/Group | Age Group 1: Patients Aged 3 to 23 Months | Age Group 2: Patients Aged 28 Days to Less Than 3 Months | Age Group 3: Patients Aged From Birth to 27 Days (Term Newborns)
Number analyzed (Participants) | 33 | 2 | 0
mg/L | 109.4 (22.4) | 116.2 (13.3) |

7. Primary Outcome: Clearance
Description: Individual predicted final model parameter scaled by body weight
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L/h/kg
Arm/Group | Age Group 1: Patients Aged 3 to 23 Months | Age Group 2: Patients Aged 28 Days to Less Than 3 Months | Age Group 3: Patients Aged From Birth to 27 Days (Term Newborns)
Number analyzed (Participants) | 33 | 2 | 0
L/h/kg | 0.128 (0.035) | 0.097 (0.004) |

8. Primary Outcome: Central Volume of Distribution (V1)
Description: Individual predicted final model parameter scaled by body weight
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L/kg
Arm/Group | Age Group 1: Patients Aged 3 to 23 Months | Age Group 2: Patients Aged 28 Days to Less Than 3 Months | Age Group 3: Patients Aged From Birth to 27 Days (Term Newborns)
Number analyzed (Participants) | 33 | 2 | 0
L/kg | 0.176 (0.033) | 0.214 (0.03) |

9. Primary Outcome: Inter-compartment Clearance (Q)
Description: Individual predicted final model parameter scaled by body weight
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L/h/kg
Arm/Group | Age Group 1: Patients Aged 3 to 23 Months | Age Group 2: Patients Aged 28 Days to Less Than 3 Months | Age Group 3: Patients Aged From Birth to 27 Days (Term Newborns)
Number analyzed (Participants) | 33 | 2 | 0
L/h/kg | 0.099 (0.025) | 0.123 (0.029) |

10. Primary Outcome: Peripheral Volume of Distribution (V2)
Description: Individual predicted final model parameter scaled by body weight
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L/kg
Arm/Group | Age Group 1: Patients Aged 3 to 23 Months | Age Group 2: Patients Aged 28 Days to Less Than 3 Months | Age Group 3: Patients Aged From Birth to 27 Days (Term Newborns)
Number analyzed (Participants) | 33 | 2 | 0
L/kg | 0.066 (0.014) | 0.066 (0.003) |

ADVERSE EVENTS:
Time Frame: Adverse events (AE) occurring from the beginning of patient's participation in the trial (Informed Consent Form signature) until the end of the participation (up to 3 months following gadopiclenol administration).
Description: Safety set population (all patients who received one administration of gadopiclenol) was used for safety evaluation. Treatment emergent AEs (AEs occurring after gadopiclenol administration) were listed below.
Arm/Group | Age Group 1: Patients Aged 3 to 23 Months | Age Group 2: Patients Aged 28 Days to Less Than 3 Months | Age Group 3: Patients Aged From Birth to 27 Days (Term Newborns)
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/2 | 0/1
Serious Adverse Events (participants affected / at risk) | 8/33 | 0/2 | 0/1
Other Adverse Events (participants affected / at risk) | 13/33 | 2/2 | 0/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Age Group 1: Patients Aged 3 to 23 Months (N=33) | Age Group 2: Patients Aged 28 Days to Less Than 3 Months (N=2) | Age Group 3: Patients Aged From Birth to 27 Days (Term Newborns) (N=1)
Feeding Disorder (Metabolism and nutrition disorders) | 1 (1) | 0 | 0 — Feeding Difficulties
Tumour Excision (Surgical and medical procedures) | 1 (1) | 0 | 0 — Tumour Resection For Suprasellar Optic Glioma
Pyrexia (General disorders) | 1 (1) | 0 | 0 — Central Fever
Microcytic Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 | 0 — Microcytic Anemia
Gastroenteritis Norovirus (Infections and infestations) | 1 (1) | 0 | 0 — Gastroenteritis - Norovirus
Pneumonia Parainfluenzae Viral (Infections and infestations) | 1 (1) | 0 | 0 — Hospitalization On Intensive Care Unit - Respiratory Failure, Pneumonia - Hpiv-3 Virus
Bronchitis (Infections and infestations) | 1 (1) | 0 | 0 — Severe Upper Respiratory Tract Infection With Severe Bronchitis
Cerebral Cyst (Nervous system disorders) | 1 (1) | 0 | 0 — Cerebral Sella Turcic Cyst Growth
Intracranial Pressure Increased (Nervous system disorders) | 1 (1) | 0 | 0 — Intercranial Hypertension
Device Malfunction (Product Issues) | 1 (1) | 0 | 0 — Disfunction Of Ventriculoperitoneal Shunt System
Renal Failure (Renal and urinary disorders) | 1 (1) | 0 | 0 — Worsening Of Pre-Existing Renal Failure
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Age Group 1: Patients Aged 3 to 23 Months (N=33) | Age Group 2: Patients Aged 28 Days to Less Than 3 Months (N=2) | Age Group 3: Patients Aged From Birth to 27 Days (Term Newborns) (N=1)
Viral Upper Respiratory Tract Infection (Infections and infestations) | 1 (1) | 0 | 0 — Upper Respiratory Viral Infection
Conjunctivitis (Infections and infestations) | 1 (1) | 0 | 0
Paronychia (Infections and infestations) | 1 (1) | 0 | 0 — Paronychia On The Toes
Hand-Foot-And-Mouth Disease (Infections and infestations) | 1 (1) | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 (1) | 0
Vomiting (Gastrointestinal disorders) | 5 (5) | 0 | 0
Anxiety (Psychiatric disorders) | 1 (1) | 0 | 0 — Anxiety
Choking (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 | 0 — Choke On Saliva
Upper Respiratory Tract Infection (Infections and infestations) | 1 (1) | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 | 0 — Light Redness Of Cheecks And Tip Of The Nose
Astigmatism (Eye disorders) | 1 (1) | 0 | 0
Myopia (Eye disorders) | 1 (1) | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 | 0 — Rash On Face
Nausea (Gastrointestinal disorders) | 1 (1) | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 | 0 — Runny Nose
White Blood Cell Count Increased (Investigations) | 1 (1) | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 | 0 — Nasal Mild Congestion
Respiratory Tract Infection Viral (Infections and infestations) | 1 (1) | 0 | 0 — Respiratory Tract Viral Illness Infection
Anaphylactic Reaction (Immune system disorders) | 1 (1) | 0 | 0 — Peanut Induced Anaphylaxis
Aspartate Aminotransferase Increased (Investigations) | 0 (0) | 1 (1) | 0
Serum Ferritin Increased (Investigations) | 0 (0) | 1 (1) | 0

LIMITATIONS AND CAVEATS:
Due to incomplete recruitment in study GDX-44-015, with only 2 patients aged 28-89 days and none aged less than 28 days who could be included in the popPK analysis, exposure in these groups was only obtained by simulation using the final model.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-10-09): https://cdn.clinicaltrials.gov/large-docs/84/NCT05590884/Prot_000.pdf
  • Statistical Analysis Plan (2024-10-29): https://cdn.clinicaltrials.gov/large-docs/84/NCT05590884/SAP_001.pdf